CLINICAL TRIAL: NCT01893801
Title: A Phase 1b/2 Pilot Trial of Nab-Paclitaxel Plus Cisplatin Plus Gemcitabine (Nabplagem) in Patients With Previously Untreated Metastatic Pancreatic Ductal Adenocarcinoma (PDA)
Brief Title: Nab-Pac+Cis+Gem in Pts w Previously Untreated Metastatic PDA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pancreatic Cancer Research Team (Other)
Collaborators: Translational Genomics Research Institute (Other); Honor Health - Clinical Trials (Unknown); Cancer Research and Biostatistics Clinical Trials Consortium (Network)
Responsible Party: Principal Investigator, Gayle Jameson, Lead Principal Investigator, Pancreatic Cancer Research Team
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCRT 12-001
Record Dates: First submitted 2013-07-02; First posted 2013-07-09 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Stage IV Pancreatic Cancer
Keywords: pancreatic cancer; pancreatic adenocarcinoma; Stage IV pancreatic cancer; pancreas; pancreatic
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nab-paclitaxel+Cisplatin+gemcitabine (Experimental): This is a phase Ib/II open-label, pilot study evaluating the preliminary efficacy and safety of nab-paclitaxel 125mb/m2, cisplatin 25mg/m2, and gemcitabine 1000mg/m2, all administered intravenously (IV) on Days 1 and 8 every 21 days until development of toxicity that is unacceptable in the opinion of the patient or the Investigator or upon disease progression.
  Interventions: Drug: nab-paclitaxel; Drug: Cisplatin; Drug: gemcitabine

INTERVENTIONS:
Drug: nab-paclitaxel — 25 mg/m2 given intravenously (IV) on days 1 and 8 of a 21 day cycle
  Other Names: Abraxane
Drug: Cisplatin — 25mg/m2 (or 50mg/m2) given intravenously (IV) on days 1 and 8 of a 21 day cycle
  Other Names: cisplatinum; cis-diamminedichloroplatinum; CDDP
Drug: gemcitabine — 1000mg/m2 given intravenously (IV) on days 1 and 8 of a 21 day cycle
  Other Names: Gemzar

SUMMARY:
The primary objective of this study is to determine the efficacy of nab-paclitaxel plus cisplatin plus gemcitabine for patients with metastatic pancreatic ductal adenocarcinoma (PDA).

DETAILED DESCRIPTION:
This is a phase 1b/2 open-label pilot study evaluating the preliminary efficacy and safety of nab-paclitaxel, cisplatin, and gemcitabine in patients with metastatic pancreatic ductal adenocarcinoma.

An individual cycle of therapy will be defined as Days 1 and 8 every 21 days. Multiple cycles may be administered until the patient is withdrawn from therapy.

Overall response rates as well as individual categories of response (complete response-CR, partial response-PR, stable disease-SD and progressive disease-PD) will be determined using RECIST 1.1. Time-to-event endpoints, including progression free survival (PFS) and OS (overall survival) will be assessed using the Kaplan-Meier method. Evaluation of stable disease at 9 weeks will also be assessed. Toxicity (adverse events) will be recorded using the NCI CTCAE (v4.0, May 2009).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years of age; male or female.
* Histologically or cytologically confirmed metastatic pancreatic ductal adenocarcinoma.
* Capable of providing informed consent and complying with trial procedures.
* Karnofsky Performance Status (KPS) of >/=70%.
* Life expectancy >/=12 weeks.
* Measurable tumor lesions according to RECIST 1.1 criteria.
* Women must not be able to become pregnant (e.g. post-menopausal for at least 1 year, surgically sterile, or practicing adequate birth control methods) for the duration of the study. Women of child bearing potential must have a negative serum or urine pregnancy test at the Screening Visit and be non-lactating. Both male and female patients of reproductive potential must agree to use a reliable method of birth control during the study.

Exclusion Criteria:

* Patients must have received no previous radiotherapy, surgery, chemotherapy or investigational therapy for the treatment of metastatic disease. Prior treatments in the adjuvant setting with gemcitabine and/or 5-FU or gemcitabine administered as a radiation sensitizer are allowed, provided at least 6 months have elapsed since completion of the last dose and no lingering toxicities are present.
* Palliative surgery and/or radiation treatment less than 4 weeks prior to initiation of study treatment.
* Exposure to any investigational agent within 4 weeks prior to initiation of study treatment.
* Evidence of central nervous system (CNS) metastasis (negative imaging study, if clinically indicated, within 4 weeks of Screening Visit).
* History of other malignancies (except cured basal cell carcinoma, superficial bladder cancer or carcinoma in situ of the cervix) unless documented free of cancer for >/= 5 years.
* Laboratory values: Screening serum creatinine > upper limits of normal (ULN); total bilirubin > ULN: alanine aminotransferase (ALT) and AST >/= 2.5 ULN or >/= 5.0 x ULN if liver metastases are present; absolute neutrophil count < 1,500/mm3, platelet concentration < 100,00/mm3, hematocrit level < 27% for females or < 30% for males, or coagulation tests (prothrombin time [PT], partial thromboplastin time [PTT], International Normalized Ratio [INR]) > 1.5 x ULN unless on therapeutic doses of warfarin.
* current, serious, clinically significant cardiac arrhythmias as determined by the Investigator.
* History of HIV infection.
* Active, clinically significant serious infection requiring treatment with antibiotics, anti-virals or anti-fungals.
* Major surgery within 4 weeks prior to initiation of study treatment. Any condition that might interfere with the patient's participation in the study or in the evaluation of the study results.
* Any condition that is unstable and could jeopardize the patient's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-05; Primary Completion 2016-04 (Actual); Study Completion 2017-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gayle S Jameson, MSN ACNP-BC, Principal Investigator — Scottsdale Health Care
Locations (3):
- United States (3):
  - Scottsdale Health Care, Scottsdale, Arizona
  - Rutgers - Cancer Institute of New Jersey (CINJ), New Brunswick, New Jersey
  - Vita Medical Associates, PC, Bethlehem, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Von Hoff DD, Ramanathan RK, Borad MJ, Laheru DA, Smith LS, Wood TE, Korn RL, Desai N, Trieu V, Iglesias JL, Zhang H, Soon-Shiong P, Shi T, Rajeshkumar NV, Maitra A, Hidalgo M. Gemcitabine plus nab-paclitaxel is an active regimen in patients with advanced pancreatic cancer: a phase I/II trial. J Clin Oncol. 2011 Dec 1;29(34):4548-54. doi: 10.1200/JCO.2011.36.5742. Epub 2011 Oct 3. PMID 21969517
- [Background] 2013 Gastrointestinal Cancers Symposium. Abstract LBA148. Presented January 25, 2013
- [Derived] Jameson GS, Borazanci E, Babiker HM, Poplin E, Niewiarowska AA, Gordon MS, Barrett MT, Rosenthal A, Stoll-D'Astice A, Crowley J, Shemanski L, Korn RL, Ansaldo K, Lebron L, Ramanathan RK, Von Hoff DD. Response Rate Following Albumin-Bound Paclitaxel Plus Gemcitabine Plus Cisplatin Treatment Among Patients With Advanced Pancreatic Cancer: A Phase 1b/2 Pilot Clinical Trial. JAMA Oncol. 2020 Jan 1;6(1):125-132. doi: 10.1001/jamaoncol.2019.3394. PMID 31580386
- See also: Additional information about the Pancreatic Cancer Research Team (PCRT) — http://www.pcrt.org
- See also: Non-profit Organization — http://www.tgen.org
- See also: Related link — http://www.td2inc.com
- See also: Non-profit organization for pancreatic cancer research — http://www.seenamagowitzfoundation.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nab-Paclitaxel+Cisplatin+Gemcitabine
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nab-Paclitaxel+Cisplatin+Gemcitabine
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (7.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
CA19-9 Status at Baseline [Count of Participants; unit: Participants]
  Abnormal | 19
  Normal | 6
CEA Status at Baseline (if CA19-9 Normal at Baseline) [Count of Participants; unit: Participants] — Population: Of the 6 patients with normal CA19-9 level at baseline, 4 (66.7%) had baseline CEA data available.
  Participants
    number analyzed (Participants) | 4
    Abnormal | 2
    Normal | 2
CA125 Status at Baseline (if CA19-9 Normal at Baseline) [Count of Participants; unit: Participants] — Population: Of the 6 patients with normal CA19-9 level at baseline, 4 (66.7%) had baseline CA125 data available.
  Participants
    number analyzed (Participants) | 4
    Abnormal | 2
    Normal | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: The primary objectives of this study is to pursue treatment of 25 individual patients with previously untreated metastatic pancreatic ductal adenocarcinoma (PDA) to evaluate:
  Complete response rate as defined by computed tomography (CT) scan using RECIST 1.1 criteria and CA 19-9 (or CA 125, or CEA if not expressers of CA 19-9) down to normal limits (from at least > 2x ULN). We expect to accomplish this in > or = to 5% of patients. When a complete response (CR) is documented, a confirmatory PET scan will be obtained.
  If 1 or more of 10 patients demonstrate a complete response (CR), study will continue to enroll to a total of 25 patients.
  If intolerable adverse events or no clinical benefit are noted in the first 6 patients, study will discontinue enrollment.
Time Frame: 1 yr.
Population: Best Response on study was assessed for patients with at least one evaluation for response while evaluable during the study. One patient achieved CR 32 days after the last dose on therapy and had a best response of PR prior to this assessment. The patient is identified as having a best response of CR in this table.
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-Paclitaxel+Cisplatin+Gemcitabine
Number analyzed (Participants) | 24
Participants
  CR | 2
  PR | 15
  SD | 4
  PD | 3
  N/A | 0

2. Secondary Outcome: Treatment-Related Toxicities
Description: Frequency of treatment-related toxicities
Time Frame: Over the course of the subjects' treatment on study, approx 1 year
Population: All patients on study were evaluated for maximum grade of treatment-related toxicity.
Measure: Count of Participants; unit: Participants
Groups:
- Nab-Pac+Cis+Gem: Nab-Paclitaxel+Cisplatin+Gemcitabine
Arm/Group | Nab-Pac+Cis+Gem
Number analyzed (Participants) | 25
Participants
  Maximum Grade 3 Treatment-Related Adverse Event | 12
  Maximum Grade 4 Treatment-Related Adverse Event | 9
  Maximum Grade 5 Treatment-Related Adverse Event | 1
  No Grade 3-5 Treatment-Related Adverse Event | 3

3. Secondary Outcome: Percentage Change in CA 19-9
Description: Percentage change in CA 19-9 from baseline values
Time Frame: Over the course of the subjects' treatment on study, approx 1 year
Population: All patients with a non-zero CA 19-9 measurement at baseline and at least one CA 19-9 measurement on-study were evaluated for percentage change of CA19-9. Of the 25 patients on study, 22 met the criteria for analysis (one had baseline CA 19-9 of zero; two had no post-baseline CA 19-9 measurements).
Measure: Mean (Standard Deviation); unit: percentage change CA 19-9 from baseline
Arm/Group | Nab-Pac+Cis+Gem
Number analyzed (Participants) | 22
percentage change CA 19-9 from baseline | -47.7 (77.13)

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from study enrollment until death from any cause.
Time Frame: Over the course of the subjects' treatment and participation in study, approx 18 mos
Population: All patients were evaluated for overall survival.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Nab-Pac+Cis+Gem: This is a Phase Ib/II open-label, pilot study evaluating the preliminary efficacy and safety of Nab-Paclitaxel 125mb/m2, Cisplatin 25mg/m2, and Gemcitabine 1000mg/m2, all administered intravenously (IV) on Days 1 and 8 every 21 days until development of toxicity that is unacceptable in the opinion of the patient or the Investigator or upon disease progression.
  Nab-Paclitaxel: 25 mg/m2 given intravenously (IV) on days 1 and 8 of a 21 day cycle
  Cisplatin: 25mg/m2 (or 50mg/m2) given intravenously (IV) on days 1 and 8 of a 21 day cycle
  Gemcitabine: 1000mg/m2 given intravenously (IV) on days 1 and 8 of a 21 day cycle
Arm/Group | Nab-Pac+Cis+Gem
Number analyzed (Participants) | 25
months | 16.4 [10.2 to 25.3]

5. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival is defined as the time from study enrollment until the first documented tumor progression (using RECIST 1.1 criteria) or death from any cause.
Time Frame: Over the course of the subjects' treatment and participation in study, approx 18 mos
Population: All patients were evaluated for progression-free survival.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-Pac+Cis+Gem
Number analyzed (Participants) | 25
months | 10.1 [6.0 to 12.5]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the period starting with initial dose of study drug and ending at the time the patient went off study or 30 days after the patient's last dose of study drug, whichever was later.
Description: The definitions of adverse event and serious adverse event for this study match the definitions from clinicaltrials.gov.
Arm/Group | Nab-Paclitaxel+Cisplatin+Gemcitabine
All-Cause Mortality (participants affected / at risk) | 21/25
Serious Adverse Events (participants affected / at risk) | 12/25
Other Adverse Events (participants affected / at risk) | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-Paclitaxel+Cisplatin+Gemcitabine (N=25)
Acute cryptosporidiosis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Anemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 2
Platelet count decreased (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Stroke (Nervous system disorders) | 2
Cardiac arrest (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-Paclitaxel+Cisplatin+Gemcitabine (N=25)
Platelet count decreased (Investigations) | 18
Neutrophil count decreased (Investigations) | 6
White blood cell decreased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 1
Lymphocyte count increased (Investigations) | 1
Anemia (Blood and lymphatic system disorders) | 7
Lung infection (Infections and infestations) | 1
Anorectal infection (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No